CLINICAL TRIAL: NCT02580227
Title: The Effect of Preoperative Tranexamic Acid on Blood Loss and Transfusion Rates in Intertrochanteric and Subtrochanteric Femur Fractures.
Brief Title: Tranexamic Acid in Intertrochanteric and Subtrochanteric Femur Fractures
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Good Samaritan Regional Medical Center, Oregon (Other)
Responsible Party: Principal Investigator, Stefan Yakel, Orthopedic Resident, Good Samaritan Regional Medical Center, Oregon
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 15-021
Record Dates: First submitted 2015-10-05; First posted 2015-10-20 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Hip Fractures; Surgical Blood Loss
Keywords: Tranexamic Acid; Blood Transfusions
MeSH Terms: conditions — Hip Fractures; Blood Loss, Surgical | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tranexamic Acid (Active Comparator): Patients will be randomized 1:1 onto active TXA arm, or placebo arm.
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): Patients will be randomized 1:1 onto active TXA arm, or placebo arm.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — All subjects will be given 1g of TXA in 100cc normal saline, or placebo of 100cc normal saline at time of admission, after consent is given.
  Arms: Tranexamic Acid
Other: Placebo — All subjects will be given 1g of TXA in 100cc normal saline, or placebo of 100cc normal saline at time of admission, after consent is given.
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the effect of Tranexamic Acid (TXA) on blood loss and need for perioperative blood transfusion following intertrochanteric and subtrochanteric femur fractures. TXA is a antifibrinolytic medication that prevents the breakdown of blood clots by inhibiting the activation of plasminogen to plasmin in the coagulation cascade. Our hypothesis is that by providing TXA at the time of hospital admission it will decrease the amount of preoperative and intraoperative bleeding thereby leading to a decreased need for post-operative transfusion. This a double blinded, placebo controlled, therapeutic trial in which half of patients will be randomized to receive TXA at the time of hospital admission and half of patients will receive a placebo.

DETAILED DESCRIPTION:
Tranexamic Acid has a long and proven history of clinical safety and effectiveness in the Orthopaedic literature. Its use in perioperative blood management in total joint arthroplasty is wide spread and is quickly becoming a standard of care. However, evidence on the effectiveness of TXA in lower extremity fracture care is more limited. There is a logical expectation that the use of TXA in lower extremity fracture care will provide a similar benefit in minimizing blood loss and reducing transfusion requirements, based on TXA's success in total joint arthroplasty, however this has not yet been validated in the literature. This study will seek to evaluate the effectiveness of TXA in perioperative blood management within a subset of lower extremity fracture, specifically intertrochanteric femur fractures. Hip fractures represent a common orthopedic injury in a fragile patient population that often necessitates post-operative blood transfusion thereby putting the patient at additional risk of complications. Intertrochanteric femur fractures have an increased risk of post-operative blood transfusion when compared to femoral neck fractures. It is presumed that the difference in blood loss between these two fracture types is caused by increased pre-operative bleeding of intertrochanteric fractures secondary to the extracapsular nature of the fracture, as opposed to a tamponade effect that occurs with intracapsular femoral neck fractures. It can therefore be expected that the use of TXA in intertrochanteric femur fractures will decrease perioperative bleeding leading to a decrease in total blood loss and a decrease in transfusion rates.

Limited research has shown that TXA is effective in reducing perioperative blood loss in hip fracture when compared to placebo, but not as effectively as when used in joint arthroplasty. One explanation for this difference is that TXA is circulating at the time of iatrogenic fracture in total joint arthroplasty or given shortly after, whereas intraoperative TXA administration in hip fractures usually doesn't occur until 6-48 hours after the initial injury. Administering TXA at the time of hospital admission in intertrochanteric femur fracture allows the drug time to decrease blood loss resulting from the fracture as well as the subsequent surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients sustaining a closed intertrochanteric femur fracture presenting to the Good Samaritan Regional Medical Center.
* Patients who are willing and able to consent to participate in the study
* >18 years of age

Exclusion Criteria:

* Patients with an allergy to tranexamic acid.
* History of thromboembolic event (pulmonary embolism, cerebral vascular accident, deep venous thrombosis),
* History of renal impairment (Cr > 1.5 or glomerular filtration rate < 30)
* Coronary stents
* History of hypercoagulability (Factor V Leiden, protein C/S deficiency, prothrombin gene mutation, anti-thrombin deficiency, anti-phospholipid antibody syndrome, lupus anticoagulant).
* Color blindness
* Subarachnoid hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-08 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Perioperative Blood Loss | Admission to discharge, 3-4 days on average.
  Perioperative blood loss measured by serial hemoglobin and hematocrit
Blood Transfusion Rates | Admission to discharge, 3-4 days on average.

OTHER OUTCOMES:
Calculated Blood Loss | Admission to discharge, 3-4 days on average.
Length of Stay | Admission to discharge, 3-4 days on average.
Myocardial Infarction | Admission to discharge, 3-4 days on average.
Deep Venous Thrombosis | Admission to discharge, 3-4 days on average.
Pulmonary Embolism | Admission to discharge, 3-4 days on average.
Cerebrovascular Accident | Admission to discharge, 3-4 days on average.
Surgical Site Infection Rate | Admission to discharge, 3-4 days on average.

CONTACTS AND LOCATIONS:
Locations (1):
- Good Samaritan Hospital Corvallis, Corvallis, Oregon, United States

REFERENCES:
- [Result] Desai SJ, Wood KS, Marsh J, Bryant D, Abdo H, Lawendy AR, Sanders DW. Factors affecting transfusion requirement after hip fracture: can we reduce the need for blood? Can J Surg. 2014 Oct;57(5):342-8. doi: 10.1503/cjs.030413. PMID 25265109
- [Result] Kadar A, Chechik O, Steinberg E, Reider E, Sternheim A. Predicting the need for blood transfusion in patients with hip fractures. Int Orthop. 2013 Apr;37(4):693-700. doi: 10.1007/s00264-013-1795-7. Epub 2013 Feb 5. PMID 23381612
- [Result] Zufferey PJ, Miquet M, Quenet S, Martin P, Adam P, Albaladejo P, Mismetti P, Molliex S; tranexamic acid in hip-fracture surgery (THIF) study. Tranexamic acid in hip fracture surgery: a randomized controlled trial. Br J Anaesth. 2010 Jan;104(1):23-30. doi: 10.1093/bja/aep314. PMID 19926634
- [Result] Vijay BS, Bedi V, Mitra S, Das B. Role of tranexamic acid in reducing postoperative blood loss and transfusion requirement in patients undergoing hip and femoral surgeries. Saudi J Anaesth. 2013 Jan;7(1):29-32. doi: 10.4103/1658-354X.109803. PMID 23717228